CLINICAL TRIAL: NCT06229262
Title: Immune and Cognitive Benefits of Mango Intake in Young Adults: A Randomized Trial
Brief Title: Immune and Cognitive Benefits of Mango Intake in Young Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Collaborators: National Mango Board (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 5230334
Record Dates: First submitted 2024-01-19; First posted 2024-01-29 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Cognition; Immunity
Keywords: Mango; Immunity; cognition

STUDY DESIGN:
Intervention Model Description: this will be a12 week, parallel study , free living with college going young adults aged 18-30 years
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator and outcome assessor will not be aware of which participant is in which arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mango Group (Active Comparator): Participants in the Mango group will consume 1.5 cups of mangos for 12 weeks
  Interventions: Dietary Supplement: Mango group
- control group (No Intervention): The control group will receive no dietary intervention. they will follow usual diet and abstain from eating mangos

INTERVENTIONS:
Dietary Supplement: Mango group — Participants will consume 1.5 cups of mangos per day for 12 weeks.
  Arms: Mango Group

SUMMARY:
The main objectives of our proposed study are to determine the effects of mango consumption on immune and cognitive functions in free-living college going young adults aged 18-30 years

DETAILED DESCRIPTION:
The main objectives of our proposed study are to determine the effects of mango consumption on immune and cognitive functions in free-living college going young adults aged 18-30. To accomplish these objectives, a randomized controlled, parallel design study is proposed with two groups consuming their habitual diet, but with one (Mango group) receiving 1.5 servings of mango/day and the other (Control group) abstaining from eating any mango for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female college students aged 18-30 years

Exclusion Criteria:

* known intolerance or allergy to mangos
* regular intake of mangos and/or fruits of a similar nutritional content such as peach, nectarine, papaya, apricot and cantaloupe
* using cognition and/or immune-boosting supplements or vitamins
* recent exposure to antibiotics and corticoids
* uncontrolled chronic diseases and mental illnesses, clinical depression, and immunocompromised state

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Changes in lymphocyte populations | baseline to 12 weeks
  Immunophenotyping will be performed by flow cytometry to measure the number of T helper, T cytotoxic, Naive and memory cells and B cells
Changes in Lymphocyte activity | baseline to 12 weeks
  The production of lymphocytes will be measured in the supernatant using enzyme linked immunosorbent assay (ELISA)
Changes in cytokine production | baseline to 12 weeks
  The cytokines produced due to lymphocyte activity will be measured in the supernatant using enzyme linked immunosorbent assay (ELISA)
Changes in serum inflammatory cytokine concentration | baseline to 12 weeks
  changes in the concentrations of the inflammatory cytokines will be performed on serum using enzyme linked immunoassay (ELISA) will include hs-CRP, interleukin (IL)-1B, IL-6, TNF a, IL-10, IL-2, IFN-γ, E-selectin,
changes from baseline in global cognitive composite score | baseline to 12 weeks
  The composite score will be calculated using the scores from the tests listed below. Scores will be calculated with the standardized scores of each test as the score of each participant minus the group mean and divide by its standard deviation. The composite score is the mean of the standardized scores. the 5 tests are: Rey Auditory Verbal Learning Test (RAVLT), Brief Visuospatial Memory Test, Digit Span, FAS Word Fluency, Symbol Digit Modalities Test
Change in serum brain-derived neurotrophic factor (pg/mL) | baseline to 12 weeks
  changes in serum brain-derived neurotrophic factor (pg/mL) assessed by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Sujatha Rajaram, PhD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University School of Public Health, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No